CLINICAL TRIAL: NCT01843413
Title: Dose Escalation for Larger Brain Metastases: Phase I/II Study
Brief Title: Stereotactic Radiosurgery in Treating Patients With Large Brain Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8312
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Tumors Metastatic to Brain; Unspecified Adult Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery; Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: Dose escalation for radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (SRS) (Experimental): Patients undergo SRS guided by CT and MRI.
  Interventions: Radiation: stereotactic radiosurgery; Procedure: quality-of-life assessment; Procedure: cognitive assessment

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Undergo SRS
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: cognitive assessment — Ancillary studies

SUMMARY:
This phase I/II trial studies the side effects and the best dose of stereotactic radiosurgery and to see how well it works in treating patients with large brain metastases. Radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the incidence of acute and long-term toxicities with increasing dose of stereotactic radiosurgery (SRS). (Phase I) II. To determine if local control may be improved with increasing doses of SRS. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the risk of acute and long-term toxicity with increasing dose of SRS. (Phase II) II. To determine if there is increased neurocognitive toxicity with increased dose of SRS.

III. To determine the rate of radiation necrosis/steroid dependency. IV. To determine if quality of life is affected more by tumor recurrence versus radiation necrosis. This includes assessment of progression free survival, overall survival, local failure, and number of patients who receive bevacizumab, laser interstitial thermal therapy, or surgery for presumed radiation necrosis.

OUTLINE: This is a phase I dose-escalation study followed by a phase II study.

Patients undergo SRS guided by computer tomography (CT) and magnetic resonance imaging (MRI).

After completion of treatment, patients are followed up at 1-2, 3, 6, 9, and 12 months, every 3 months for 2 years, and then every 4 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing SRS for brain metastases
* Lesions to be treated under this protocol must be > 2 cm, but =< 4.0 cm in diameter
* Patients may have had prior therapy including:

  * Whole brain radiation therapy (WBRT) > 3 months ago
  * SRS to other brain metastases
* Patients with newly diagnosed brain metastases are eligible as long as they are not planned for WBRT upfront
* Any primary is eligible with exception of small cell lung cancer, lymphoma, and germ cell histologies
* Patient must be able to provide written informed consent

Exclusion Criteria:

* Patients receiving SRS to resection bed
* Planned concurrent WBRT
* Leptomeningeal metastases
* Small cell lung cancer, lymphoma, and germ cell histologies
* Inability to participate in study activities due to physical or mental limitations
* Inability or unwillingness to return for all the required follow-up visits
* Conformality index 2.0 or less cannot be achieved, or homogeneity index is > 2.0
* Unable to deliver 10 Gray (Gy) or less to optic nerve/chiasm
* Brainstem location is excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose based on the incidence of dose-limiting toxicity (DLT) defined as any grade III or IV toxicity as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | Up to 4 months
Response associated with increased dose of SRS as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) (Phase II) | Up to 2 years

SECONDARY OUTCOMES:
Incidence of adverse events as assessed by CTCAE version 4.0 (Phase II) | Up to 2 years
  Toxicity will be summarized as frequencies and percentages with a corresponding exact 95% confidence interval.
Quality of life (QOL) as assessed by the Functional Assessment of Cancer Therapy-Brain (FACT-BR) and the European Organization for Research and Treatment (EORTC)- Quality of Life Questionnaire Core 30 (QLQ30) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Chao, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States